CLINICAL TRIAL: NCT02312024
Title: International Registry on the Use of the CytoSorb®-Adsorber in ICU Patients
Brief Title: International Registry on the Use of the CytoSorb Adsorber
Acronym: CytoSorb
Status: Completed | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: University Hospital Goettingen (Other)
Responsible Party: Sponsor
Other Study IDs: JenaUH
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2024-10-23 (Actual); Status verified 2019-12

CONDITIONS: Sepsis; Need of Cardiac Surgery
Keywords: CytoSorb adsorber; sepsis; cytokines; hemofiltration; hemadsorption; inflammation
MeSH Terms: conditions — Sepsis; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with severe sepsis/septic shock: Use of CytoSorb adsorber in patients with severe sepsis/septic shock
  Interventions: Device: Use of CytoSorb adsorber
- Cardiac surgery with CPB: preemptive use: Use of CytoSorb adsorber in patients with cardiac surgery with CPB: preemptive use
- Cardiac surgery with CPB: postop. use: Use of CytoSorb adsorber in patients with cardiac surgery with CPB: postoperative use
- Patients with other indications: Use of CytoSorb adsorber in patients with other indications
  Interventions: Device: Use of CytoSorb adsorber

INTERVENTIONS:
Device: Use of CytoSorb adsorber — Use of CytoSorb adsorber either in patients with severe sepsis/septic shock or with cardiac surgery with CPB or in other patients.
  Groups: Patients with other indications; Patients with severe sepsis/septic shock

SUMMARY:
Registry on the use of the CytoSorb® adsorber in ICU patients.

DETAILED DESCRIPTION:
The aim of this registry is to record the use of CytoSorb® under real life conditions in as many cases as possible (preferably all or, at least, in a representative sample). All CytoSorb® applications in different clinical settings and in all patients who are treated with this technology in Germany, Austria and Switzerland (target population) are planned to be included.

The objectives of the registry are collection of real-life data on a broad scale, their centralized, structured and comprehensive documentation, and a controlled data exchange. The gathered information will be used to augment the knowledge on the clinical efficacy of the technology, to optimize the quality of its therapeutic application, and to identify and promptly handle possible complications related to the use of CytoSorb®. The registry will record all relevant information in the course of product use, e.g. diagnosis, comorbidities, course of the condition, treatment, concomitant medication and clinical laboratory parameters.

The registry will inform physicians of different medical specialties about the range of possible applications of CytoSorb® and invite them to contribute their own experiences to the registry. This is done by giving them access to their own data and to the results of periodic analyses (for contributing participants), and via publications of the results (for participants and external interested parties)

The CytoSorb® registry will provide the data base for justified and optimized decisions. An active form of data collection where data is prospectively collected by qualified staff is particularly suited for this purpose.

Registry data might help closing knowledge gaps and open practical issues. Due to the patient group's heterogeneity, the registry can identify sub-groups, assess their risk-benefit-profile and examine their safety profile. Registry data are absolutely essential for assessing a therapy's significance within the healthcare landscape.

Institutions that contribute data to the registry benefit in several ways: They will obtain a continuous retrospective feedback of their own results, their data will be periodically compared with data from other participating sites, and they will get access to regularly published analyses of the results of all participants. On the basis of these data, they can establish a quality monitoring and optimize their use of CytoSorb®.

The planned endpoints allow for a comprehensive description of CytoSorb® efficacy in terms of several indication-relevant aspects. Together with the monitoring of application safety, these data build the basis for establishing benchmarks that promote a higher treatment quality.

ELIGIBILITY:
Inclusion Criteria:

* Use of the CytoSorb® adsorber
* Age ≥ 18 years
* Signed informed consent

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing treatment with the CytoSorb® adsorber
Sampling Method: Non-Probability Sample
Enrollment: 1434 (Actual)
Dates: Start 2015-01; Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Difference between mortality predicted by scoring systems (APACHE II/SAPS II, EuroSCORE II) and actual mortality within 30 days after intervention | days

SECONDARY OUTCOMES:
- Organ function (SOFA - score-difference) | days
- Concentration of biomarkers IL-6, CRP, PCT, myoglobin, free hemoglobin | days
- Length of hospital and ICU stay (days) | days
- Duration of mechanical ventilation (days) | days
- Duration of renal replacement therapy (days) | days
- Duration of vasopressor therapy (days) | days

CONTACTS AND LOCATIONS:
Overall Officials: Frank M. Brunkhorst, Prof., Principal Investigator — Center for Clinical Studies at Jena University Hospital
Locations (19):
- Krankenhaus Hietzing, Vienna, Austria
- Germany (17):
  - Vivantes Klinikum Neukölln, Berlin
  - Evangelisches Krankenhaus, Bielefeld
  - Carl-Thiem-Klinikum, Cottbus
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Klinikum Emden, Emden
  - Kliniken Erlabrunn gGmbH, Erlabrunn
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - Greifswald University Hospital, Greifswald
  - Krankenhaus St. Elisabeth & St. Barbara, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Krankenhaus Herzberg, Elbe-Elster-Klinikum GmbH, Herzberg
  - Kliniken Maria Hilf GmbH Mönchengladbach, Mönchengladbach
  - Klinikum rechts der Isar der TU München, München
  - Klinikum Oldenburg, Oldenburg
  - University Hospital Ulm, Ulm
  - Kliniken Nordoberpfalz AG, Klinikum Weiden, Weiden
- University of Szeged, Szeged, Hungary

REFERENCES:
- [Background] Hawchar F, Tomescu D, Trager K, Joskowiak D, Kogelmann K, Soukup J, Friesecke S, Jacob D, Gummert J, Faltlhauser A, Aucella F, van Tellingen M, Malbrain MLNG, Bogdanski R, Weiss G, Herbrich A, Utzolino S, Nierhaus A, Baumann A, Hartjes A, Henzler D, Grigoryev E, Fritz H, Bach F, Schroder S, Weyland A, Gottschaldt U, Menzel M, Zachariae O, Novak R, Berden J, Haake H, Quintel M, Kloesel S, Kortgen A, Stecher S, Torti P, Nestler F, Nitsch M, Olboeter D, Muck P, Findeisen M, Bitzinger D, Krassler J, Benad M, Schott M, Schumacher U, Molnar Z, Brunkhorst FM. Hemoadsorption in the critically ill-Final results of the International CytoSorb Registry. PLoS One. 2022 Oct 25;17(10):e0274315. doi: 10.1371/journal.pone.0274315. eCollection 2022. PMID 36282800
- [Derived] Schittek GA, Zoidl P, Eichinger M, Orlob S, Simonis H, Rief M, Metnitz P, Fellinger T, Soukup J. Adsorption therapy in critically ill with septic shock and acute kidney injury: a retrospective and prospective cohort study. Ann Intensive Care. 2020 Nov 18;10(1):154. doi: 10.1186/s13613-020-00772-7. PMID 33206229
- [Derived] Friesecke S, Trager K, Schittek GA, Molnar Z, Bach F, Kogelmann K, Bogdanski R, Weyland A, Nierhaus A, Nestler F, Olboeter D, Tomescu D, Jacob D, Haake H, Grigoryev E, Nitsch M, Baumann A, Quintel M, Schott M, Kielstein JT, Meier-Hellmann A, Born F, Schumacher U, Singer M, Kellum J, Brunkhorst FM. International registry on the use of the CytoSorb(R) adsorber in ICU patients : Study protocol and preliminary results. Med Klin Intensivmed Notfmed. 2019 Nov;114(8):699-707. doi: 10.1007/s00063-017-0342-5. Epub 2017 Sep 4. PMID 28871441
- See also: Project website — http://www.cytosorb-registry.org